CLINICAL TRIAL: NCT07243314
Title: Evaluating Functional Outcomes of 3D-Printed Splints in Post-Stroke Upper Limb Recovery
Acronym: 3D-splint
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Zainab Saud Alshammari, Physical therapist, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No.: 151-2025-IRB; Not found (Other: Not found)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Stroke Rehabilitation; Hemiparesis of the Upper Limb Following Stroke
Keywords: stroke; Ischemic Stroke; Hemorrhagic Stroke; Hemiparesis; Splint; Dynamic Splint; Three-Dimensional Printing; 3D-Printed Splint; Orthosis; Task-Oriented; Traditional Dynamic Splint; Motor Function
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-Printed Dynamic Splint Group (Experimental): will wear a 3D-printed dynamic splint at least 6 hours daily
  Interventions: Device: 3D Printed splint
- Dynamic Splint Group (Active Comparator): will wear a conventional dynamic splint for at at least 6 hours
  Interventions: Device: conventional splint

INTERVENTIONS:
Device: 3D Printed splint — Patients undergo 60-minute therapy sessions 5 times per week for 4 weeks, including stretching and task-oriented training.
  Splint Protocol: A 3D-printed dynamic splint is worn during the 60-minute clinic session, plus an additional 5 hours daily on training days and 6 hours daily on non-training days
  Arms: 3D-Printed Dynamic Splint Group
Device: conventional splint — Patients undergo 60-minute therapy sessions 5 times per week for 4 weeks, including stretching and task-oriented training.
  Splint Protocol: A conventional dynamic splint is worn during the 60-minute clinic session, plus an additional 5 hours daily on training days and 6 hours daily on non-training days
  Arms: Dynamic Splint Group

SUMMARY:
This study aims to evaluate the upper limb motor recovery using a 3D-printed dynamic orthosis compared to a conventional one as part of a rehabilitation program in individuals with chronic stroke.

The main question it seeks to answer:

Which type of dynamic splint (3D-printed or traditional), combined with the task-oriented therapy program, leads to greater improvement in affected upper-limb function, patient satisfaction, and usability in stroke patients? Researchers will compare these two types of dynamic splints.

Participants will:

Receive 20 sessions of task-oriented therapy combined with either a 3D-printed dynamic splint or a traditional dynamic splint.

Visit the clinic five times a week for a period of four weeks. Undergo assessments before and after the 4-week program.

DETAILED DESCRIPTION:
Background: After a stroke, intensive motor rehabilitation is essential to improve upper limb function and independence. 3D-printed dynamic splints offer precise joint alignment, adjustable resistance, and enhanced comfort, facilitating repetitive, task-oriented practice and promoting neuroplasticity. To date, no studies have directly compared the effectiveness of 3D-printed dynamic splints with conventional dynamic splints combined with task-oriented therapy for improving upper limb function after stroke. Objectives: To evaluate the effects of 3D-printed versus conventional dynamic splints, both combined with task-oriented therapy, on upper limb motor recovery and patient satisfaction in chronic stroke patients. Methods: A randomized controlled trial will assign participants to either a 3D-printed splint + task-oriented therapy group or a conventional splint + therapy group. The intervention will last 4 weeks, with five 60-minute sessions per week, and daily splint use for 6 hours.

Inclusion Criteria: Adults ≥18 years with chronic stroke and upper limb hemiparesis, able to understand and follow instructions, MMSE ≥24, mild to moderate upper-limb spasticity, and not participating in other clinical or research studies simultaneously. Exclusion Criteria: Severe spasticity, upper limb deformities or contractures, unilateral neglect, or severe language or cognitive impairments.Outcomes: Primary outcomes: Fugl-Meyer Assessment for Upper Extremity (FMA-UE), Wolf Motor Function Test (WMFT), Box and Block Test (BBT). Secondary outcomes: Motor Activity Log (MAL), Arabic version of Stroke Impact Scale (SIS-16), and Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0).

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old.
2. Chronic stroke
3. Upper limb hemiparalysis
4. Ability to understand and follow orders and able to provide informed consent (Mini-Mental State Exam (MMSE) > 24)
5. Upper-limb mild to moderate spasticity (Modified Ashworth Scale 1+ to 3 at the wrist).
6. Not participating in other clinical or research studies at the same time

Exclusion Criteria:

1. Had deficits in language or cognitive impairments that were likely to interfere with their cooperation in the study
2. Deformity or presented with severe upper-limb contractures
3. Inability to commit to the time requirement of the protocol.
4. Unilateral neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test (WMFT) | at baseline and after intervention (4 weeks)
  The WMFT is a standardized assessment used to measure upper extremity motor ability through the performance of 17 tasks that include both functional and strength components. Rated using the 6-point scale ranging from 0 (no attempt) to 5 (normal movement). The total performance time and quality of movement are recorded, with lower scores indicating lower levels of functioning.
Fugl-Meyer Assessment Scale for Upper Extremity (FMA-UE) | at baseline and after intervention (4 weeks)
  The FMA-UE is a comprehensive quantitative measure designed to evaluate motor function, coordination, and reflex activity of the affected upper limb following stroke. It uses a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully), with a maximum score of 66 points for the upper extremity. It is considered the gold standard for assessment of upper limb motor recovery.
Box and Block Test (BBT) | at baseline and after intervention (4 weeks)
  The BBT is a validated measure of gross manual dexterity that evaluates how many 1-inch wooden blocks a participant can transfer from one compartment to another within 60 seconds using one hand. The apparatus consists of a wooden box divided into two equal sections containing 150 small cubes. The test begins with the unaffected upper limb to allow practice and establish a baseline performance. Participants are then instructed to move as many blocks as possible, one at a time, over the partition within the time limit. The score is defined as the total number of blocks successfully transferred within 60 seconds.

SECONDARY OUTCOMES:
Motor Activity Log (MAL) | at baseline and after intervention (4 weeks)
  MAL is a validated, self-reported questionnaire that assesses the real-world use of the affected upper limb during activities of daily living. It consists of two subscales: the Amount of Use (AOU) and the Quality of Movement (QOM). Each subscale contains 30 items rated on a 6-point Likert scale. For the AOU subscale, participants rate how frequently they used their affected arm, from 0 ("did not use my weaker arm") to 5 ("used my weaker arm as often as before the stroke"). For the QOM subscale, participants rate how well the affected limb assisted in the task, from 0 ("my weaker arm was not used at all for that activity") to 5 ("the ability to use my weaker arm was as good as before the stroke").
Arabic Version of Stroke Impact Scale (SIS-16) | at baseline and after intervention (4 weeks)
  The SIS-16 is a self-report tool designed to evaluate health-related quality of life among stroke survivors. It includes 16 items covering mobility, self-care, and hand function, rated on a 5-point Likert scale (1 = unable to do, 5 = not difficult at all). Higher scores represent a better level of health-related quality of life status for stroke patients.
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | Each session (5 times per week)
  QUEST 2.0 assesses user satisfaction with assistive devices and related services through 12 items divided into two subscales: device satisfaction and service satisfaction. Each item is rated on a 5-point Likert scale (1 = not satisfied at all, 5 = very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Bin Abdulaziz Humanitarian City, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- [Result] Zheng Y, Liu G, Yu L, Wang Y, Fang Y, Shen Y, Huang X, Qiao L, Yang J, Zhang Y, Hua Z. Effects of a 3D-printed orthosis compared to a low-temperature thermoplastic plate orthosis on wrist flexor spasticity in chronic hemiparetic stroke patients: a randomized controlled trial. Clin Rehabil. 2020 Feb;34(2):194-204. doi: 10.1177/0269215519885174. Epub 2019 Nov 5. PMID 31686529
- [Result] Jeon HS, Woo YK, Yi CH, Kwon OY, Jung MY, Lee YH, Hwang S, Choi BR. Effect of intensive training with a spring-assisted hand orthosis on movement smoothness in upper extremity following stroke: a pilot clinical trial. Top Stroke Rehabil. 2012 Jul-Aug;19(4):320-8. doi: 10.1310/tsr1904-320. PMID 22750961
- [Result] Andringa AS, Van de Port IG, Meijer JW. Tolerance and effectiveness of a new dynamic hand-wrist orthosis in chronic stroke patients. NeuroRehabilitation. 2013;33(2):225-31. doi: 10.3233/NRE-130949. PMID 23949058
- [Result] Yang YS, Tseng CH, Fang WC, Han IW, Huang SC. Effectiveness of a New 3D-Printed Dynamic Hand-Wrist Splint on Hand Motor Function and Spasticity in Chronic Stroke Patients. J Clin Med. 2021 Sep 30;10(19):4549. doi: 10.3390/jcm10194549. PMID 34640564
- [Result] Chen ZH, Yang YL, Lin KW, Sun PC, Chen CS. Functional Assessment of 3D-Printed Multifunction Assistive Hand Device for Chronic Stroke Patients. IEEE Trans Neural Syst Rehabil Eng. 2022;30:1261-1266. doi: 10.1109/TNSRE.2022.3173034. Epub 2022 May 17. PMID 35533167